CLINICAL TRIAL: NCT00547378
Title: Prospective, Multicenter Trial Evaluating the Safety and Efficacy of InterStim® Therapy in Subjects With Symptoms of Overactive Bladder (InSite OAB)
Brief Title: InSite for Over Active Bladder
Acronym: InSite - OAB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Protocol 1634; NCT00549094 (obsolete NCT alias)
Record Dates: First submitted 2007-10-18; First posted 2007-10-22 (Estimated); Results first posted 2017-12-12 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-11

CONDITIONS: Urinary Incontinence, Urgency-frequency; Overactive Bladder
Keywords: overactive bladder, urinary incontinence, incontinence,Urgency-frequency
MeSH Terms: conditions — Urinary Incontinence; Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): InterStim Therapy
  Interventions: Device: InterStim
- 2 (Active Comparator): Standard Medical Therapy
  Interventions: Drug: Standard Medical Therapy

INTERVENTIONS:
Device: InterStim
  Arms: 1
Drug: Standard Medical Therapy — Oxybutynin 2.5mg, 5mg Oxybutynin extended release 5 mg, 10mg, 15mg Oxybutynin transdermal 3.9mg Solifenacin 5mg, 10mg Tolterodine 1mg, 2mg Tolterodine extended release 2mg, 4mg Trospium 20mg Darifenacin extended release 7.5mg, 15mg fesoterodine Fumarate 4mg, 8mg
  Arms: 2

SUMMARY:
The purposes of this study are:

1. To provide evidence from a randomized controlled trial that InterStim Therapy provides better relief of symptoms of OAB than standard medical treatments in current use.
2. To fulfill the requirements of the FDA-mandated post-approval study of the safety of the tined lead using a minimally invasive approach.

DETAILED DESCRIPTION:
Approximately 30 million Americans meet the criteria for overactive bladder (OAB). Urinary voiding dysfunction symptoms impose a significant physical and psychosocial impact on individuals, including loss of self-esteem and a decrease in the ability to maintain an independent lifestyle. These symptoms can substantially affect a subject's daily activities.

Patients with OAB are managed with diet modification, bladder training or retraining, pelvic muscle rehabilitation, medication and biofeedback. Medications are used as the first-line therapy for urgency frequency and urinary urge incontinence.

InterStim Therapy utilizes sacral nerve stimulation and is indicated in the US for the treatment of urinary retention and the symptoms of OAB, including urinary urge incontinence and significant symptoms of urgency-frequency alone or in combination, in subjects who have failed or could not tolerate more conservative treatments.

InSite OAB Protocol 1634 consists of two phases; Phase I which is the randomized portion of the trail and Phase II the non-randomized portion.

Phase 1: A minimum of 60 subjects randomized to InterStim and a minimum of 60 subjects randomized to SMT.

Phase 2: Non-randomized, all qualified subjects will receive InterStim, approximately 297 enrolled Subjects previously enrolled in Protocol 1634 for Urinary Urge Incontinence and Protocol 1635 for Urgency-Frequency will be included in Phase I of the new Protocol 1634 of OAB.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of OAB including urinary urge incontinence or urgency-frequency
* Be male or female at least 18 years of age or older
* Be able to consent to participate by signing the Informed Consent
* Be willing and able to attend visits and comply with the study protocol including adequate operation of equipment
* Have failed or are not a candidate for more conservative treatment (e.g. pelvic floor training, biofeedback, behavioral modification)
* Have failed or could not tolerate (stopped taking medication due to lack of efficacy or intolerable side effects) at least one anticholinergic or antimuscarinic medication AND have at least one anticholinergic or antimuscarinic medication not yet attempted
* Have been on current regiment of OAB medications or have not been on any OAB medications, for at least 4 weeks prior to beginning the baseline voiding diary

Exclusion Criteria:

* Have severe or uncontrolled diabetes or diabetes with peripheral nerve involvement
* Have concomitant medical conditions which would limit the success of the study procedure
* Have skin, orthopedic or neurologic anatomical limitations that could prevent successful placement of an electrode
* Have neurological diseases such as multiple sclerosis, clinically significant peripheral neuropathy or complete spinal cord injury (e.g., paraplegia)
* Have knowledge of planned MRIs, diathermy, microwave exposure, high output ultrasonic exposure, or RF energy exposure
* Have urinary tract mechanical obstruction such as benign prostatic hypertrophy, cancer, or urethral stricture
* Have symptomatic urinary tract infection (UTI)
* Have implantable neurostimulators, pacemakers, or defibrillators
* Have primary stress incontinence or mixed incontinence where the stress component overrides the urge component
* Have had treatment of urinary symptoms with botulinum toxin therapy in the past 12 months
* Be a woman who is pregnant or planning to become pregnant or are a woman of child-bearing potential who is not using a medically-acceptable method of birth control
* Have a life expectancy of less than one year
* Have plans to enroll in another investigation device or drug trial during their participation in this trial, or currently enrolled in an investigational device or drug trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 571 (Actual)
Dates: Start 2007-10; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Siegel, MD, Study Chair — Metro Urology

REFERENCES:
- [Derived] Siegel S, Noblett K, Mangel J, Griebling TL, Sutherland SE, Bird ET, Comiter C, Culkin D, Bennett J, Zylstra S, Berg KC, Kan F, Irwin CP. Results of a prospective, randomized, multicenter study evaluating sacral neuromodulation with InterStim therapy compared to standard medical therapy at 6-months in subjects with mild symptoms of overactive bladder. Neurourol Urodyn. 2015 Mar;34(3):224-30. doi: 10.1002/nau.22544. Epub 2014 Jan 10. PMID 24415559

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty-eight centers were activated to enroll subjects. In total, 571 subjects were enrolled: 243 randomized cohort (96 excluded due to eligibility failure); 328 non-randomized cohort (102 excluded due to declined to participate; did not meet inclusion criteria and other). Subjects were enrolled between November 2007 and March 10, 2011.
Pre-assignment Details: The study has 2 cohorts. The randomized cohort included subjects who were randomized 1:1 to either InterStim Therapy (IST) or Standard Medical Therapy (SMT) and were followed for 6 months. The all implanted cohort include implanted subjects from the randomized cohort plus additional subjects enrolled after randomized cohort enrollment completion.
Groups:
- InterStim Therapy: Randomized Cohort - InterStim Therapy. This includes those subjects who were randomized to InterStim Therapy.
- Standard Medical Therapy: Randomized Cohort - Standard Medical Therapy. This includes subjects who were randomized to Standard Medical Therapy. After being followed at SMT Month 6, these subjects could choose to receive test stimulation and if successful, received full system implant.
- All Implanted/Non-Randomized Cohort: These additional subjects were not randomized. These non-randomized subjects went through test stimulation and, if successful, were implanted with the InterStim Therapy system.
Period: Randomized Cohort
Arm/Group | InterStim Therapy | Standard Medical Therapy | All Implanted/Non-Randomized Cohort
Started | 70 | 77 | 0
Month 3 | 62 (This includes IST subjects reached Month 3 visit, regardless of implant or not.) | 72 (This included SMT subjects who reached SMT Month 3 visit.) | 0
Month 6 | 59 (This includes IST subjects reached Month 6 visit, regardless of implant or not.) | 71 (This included SMT subjects who reached SMT Month 6 visit.) | 0
Completed | 59 | 71 | 0
Not Completed | 11 | 6 | 0
Not completed — Withdrawal by Subject | 7 | 5 | 0
Not completed — Death | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Other reasons | 2 | 0 | 0
Period: All Implanted Cohort
Arm/Group | InterStim Therapy | Standard Medical Therapy | All Implanted/Non-Randomized Cohort
Started (Subjects went through test stimulation in each group; if successful, received a full system implant.) | 51 (This included subjects who received full system implant after randomized to IST.) | 40 (This included SMT subjects who received full system implant after completing randomization period.) | 181 (This included subjects who received full system implant from non-randomized subjects.)
Month 3 | 51 | 39 | 178
Month 6 | 50 | 36 | 178
Month 12 | 48 | 32 | 175
Month 24 | 42 | 30 | 161
Month 36 | 42 | 29 | 146
Month 48 | 38 | 27 | 136
Month 60 | 36 | 23 | 114
Completed | 36 | 22 | 111
Not Completed | 15 | 18 | 70
Not completed — Withdrawal by Subject | 5 | 4 | 27
Not completed — Adverse Event | 4 | 10 | 17
Not completed — Lost to Follow-up | 0 | 1 | 14
Not completed — Death | 3 | 1 | 4
Not completed — Physician Decision | 0 | 2 | 6
Not completed — Site closure | 2 | 0 | 1
Not completed — Other reasons | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Randomized Cohort: InterStim Therapy: This includes those subjects who were randomized to InterStim Therapy.
- Randomized Cohort: Standard Medical Therapy: This includes subjects who were randomized to Standard Medical Therapy. After being followed at SMT Month 6, these subjects could choose to receive test stimulation and if successful, received full system implant.
- All Implanted Cohort: Non-randomized Subjects: These additional subjects were not randomized. These non-randomized subjects went through test stimulation and, if successful, were implanted with the InterStim Therapy system.
- Total: Total of all reporting groups
Arm/Group | Randomized Cohort: InterStim Therapy | Randomized Cohort: Standard Medical Therapy | All Implanted Cohort: Non-randomized Subjects | Total
Number analyzed (Participants) | 70 | 77 | 181 | 328
Age, Customized [Mean (Standard Deviation); unit: years]
  Age, years | 60.4 (14.4) | 57.1 (15.3) | 57.2 (14.1) | 57.9 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 71 | 165 | 302
  Male | 4 | 6 | 16 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 8 | 11
  Not Hispanic or Latino | 67 | 77 | 173 | 317
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 61 | 70 | 161 | 292
  Race: Black | 7 | 7 | 12 | 26
  Race: Asian/White | 1 | 0 | 0 | 1
  Race: American Indian or Alaska Native/White | 0 | 0 | 2 | 2
  Race: American Indian or Alaska Native | 0 | 0 | 1 | 1
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Race: Other | 1 | 0 | 4 | 5
Baseline Leaks/Day [Mean (Standard Deviation); unit: Leaks/Day] — Population: Leaks and voids include only those subjects who qualified for Urinary Urge Incontinence (leaks) or Urgency Frequency (voids) at baseline as demonstrated on a 3-day voiding diary demonstrating greater than or equal to 8 voids per day and/or by having a minimum of 2 involuntary leaking episodes in 72 hours. A subject could qualify for both.
  Leaks/Day
    number analyzed (Participants) | 51 | 61 | 138 | 250
    (all) | 2.4 (1.7) | 2.7 (1.9) | 3.4 (3.0) | 3.0 (2.6)
Baseline Voids/Day [Mean (Standard Deviation); unit: Voids/Day] — Population: Leaks and voids include only those subjects who qualified for Urinary Urge Incontinence (leaks) or Urgency Frequency (voids) at baseline as demonstrated on a 3-day voiding diary demonstrating greater than or equal to 8 voids per day and/or by having a minimum of 2 involuntary leaking episodes in 72 hours. A subject could qualify for both.
  Voids/Day
    number analyzed (Participants) | 45 | 50 | 134 | 229
    (all) | 11.2 (2.9) | 11.9 (4.3) | 13.1 (4.8) | 12.5 (4.5)

OUTCOME MEASURES:

1. Primary Outcome: Randomized Cohort: OAB Therapeutic Response
Description: To demonstrate that the OAB therapeutic response rate at 6 months is greater for the InterStim therapy group than for the Standard Medical Therapy group. OAB therapeutic response rate was calculated as number of subjects with OAB therapeutic response divided by number of subjects included in the analysis. OAB therapeutic response was defined as:
  * at least 50% or greater improvement in average leaks/day from baseline for subjects with urinary incontinence at baseline or
  * at least 50% improvement in average voids/day from baseline or a return to normal voiding frequency (<8 voids/day) for subjects with urgency-frequency at baseline.
Time Frame: 6 months
Population: Intent-to-Treat (ITT): an analysis that includes all randomized subjects. This was analysis in the randomized cohort.
Measure: Number; unit: percentage of participants with response
Groups:
- InterStim Therapy: Subjects who were randomized to InterStim Therapy group
- Standard Medical Therapy: Subjects who were randomized to Standard Medical Therapy group
Arm/Group | InterStim Therapy | Standard Medical Therapy
Number analyzed (Participants) | 70 | 77
percentage of participants with response | 61 | 42
Statistical Analysis 1: Comparison: InterStim Therapy vs Standard Medical Therapy; Test type: Superiority; p = 0.016, Cochran-Mantel-Haenszel; The two-sided Cochran-Mantel-Haenszel (CMH) test, stratified for center, was used to test the difference in responder rates between the 2 groups

2. Primary Outcome: All Implanted Cohort: Adverse Events Related to the Tined Lead That Require Surgery
Description: To demonstrate that the upper bound of the 95% CI for the cumulative five-year rate of adverse events related to the tined lead that require surgery is less than 0.33.
  Adverse events on or after neurostimulator implant with an etiology of lead and with an intervention of surgical intervention/revision are the event of interest.
Time Frame: 5 years
Population: This objective was analyzed in the all implanted cohort.
Measure: Number (95% Confidence Interval); unit: Cumulative probability at 5 years
Groups:
- All Implanted Cohort: The all implanted cohort included implanted subjects from the initial randomized cohort plus additional subjects enrolled in the study after the randomized cohort enrollment was complete. These additional subjects were not randomized. These non-randomized subjects went through test stimulation and, if successful, were implanted with the InterStim Therapy system. All implanted subjects were followed for 5 years.
Arm/Group | All Implanted Cohort
Number analyzed (Participants) | 272
Cumulative probability at 5 years | 0.224 [0.166 to 0.277]

3. Secondary Outcome: All Implanted Cohort: Tined Lead Migration Rate
Description: To estimate the suspected cumulative tined lead migration rate at 5 years in subjects with a full system implant. Suspected tined lead migration resulting in an adverse event of lead migration/dislodgement meets the definition of this endpoint.
Time Frame: 5 years
Population: This objective was analyzed in the all implanted cohort.
Measure: Number (95% Confidence Interval); unit: Cumulative probability at 5 years
Arm/Group | All Implanted Cohort
Number analyzed (Participants) | 272
Cumulative probability at 5 years | 0.059 [0.029 to 0.089]

4. Secondary Outcome: All Implanted Cohort: Infection Rate Associated With the Tined Lead
Description: To characterize the cumulative infection rate at 5 years associated with the tined lead in subjects with a full system implant.
Time Frame: 5 years
Population: This objective was analyzed in the all implanted cohort.
Measure: Number (95% Confidence Interval); unit: Cumulative probability at 5 years
Arm/Group | All Implanted Cohort
Number analyzed (Participants) | 272
Cumulative probability at 5 years | 0.012 [0 to 0.025]

ADVERSE EVENTS:
Time Frame: Randomization to 6 months follow-up for InterStim arm and Standard Medical Therapy arm in randomized cohort. Implant to 5-year follow up for all implanted cohort.
Description: This section presents the adverse events (regardless device related or otherwise) occurred between randomization and 6 months follow-up in the randomized cohort; and the adverse events (regardless device related or otherwise) occurred post implant through 5-year follow-up for all implanted cohort. The adverse events post implant for InterStim arm subjects in randomized cohort were also included in the adverse events summary of all implanted cohort.
Groups:
- Randomized Cohort: InterStim Therapy Group: Adverse events are summarized for those subjects randomized to the InterStim Therapy group and received full system implant (n=51). Out of 70 subjects, there are 11 subjects who were not implanted with any device component, and 8 subjects who were implanted with lead only, but no neurostimulator. These subjects were not included in this summary. For comparision purpose, adverse events are tabluated between those subjects who received InterStim therapy vs. those who were compliant with Standard Medical Therapy.
- Randomized Cohort: Standard Medical Therapy Group: Adverse events are summarized for those Subjects randomized are compliant to Standard Medical Therapy group (n=75). Out of 77 subjects, 2 subjects crossovered to InterStim Therapy group and received implant. These subjects are not included in this summary. For comparision purpose, adverse events are tabluated between those subjects who received InterStim therapy vs. those who were compliant with Standard Medical Therapy.
Arm/Group | Randomized Cohort: InterStim Therapy Group | Randomized Cohort: Standard Medical Therapy Group | All Implanted Cohort
All-Cause Mortality (participants affected / at risk) | 0/51 | 1/75 | 8/272
Serious Adverse Events (participants affected / at risk) | 5/51 | 4/75 | 107/272
Other Adverse Events (participants affected / at risk) | 29/51 | 22/75 | 217/272
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized Cohort: InterStim Therapy Group (N=51) | Randomized Cohort: Standard Medical Therapy Group (N=75) | All Implanted Cohort (N=272)
Hepatic enzyme abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 3 (4)
Sick sinus syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 3 (3)
Toe deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Vaginal cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Affective disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 4 (5)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 12 (13)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 7 (8)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 5 (12)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 5 (5)
Chest pain (General disorders) | 0 (0) | 0 (0) | 5 (6)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 4 (5)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 3 (5)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 3 (5)
Chronic obstructive airways disease exacerbated (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (5)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3)
Clostridial infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Lobar pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Asthenia (General disorders) | 0 (0) | 0 (0) | 2 (2)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Intentional misuse (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Catheter bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Escherichia sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Listeria encephalitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Meningitis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Adrenal mass (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 0 (0) | 1 (2)
Diabetes mellitus non-insulin-dependent (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Conversion disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2)
Arachnoid cyst (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebellar haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cubital tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Global amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Mononeuropathy multiplex (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Normal pressure hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (3)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Aortic disorder (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Venous insufficiency (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumoperitoneum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rectocele (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Cystitis interstitial (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Cystocele (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pregnancy (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pelvic prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Uterine enlargement (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Adenomatous polyposis coli (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Hereditary spastic paraplegia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Spondylolisthesis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Hernia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Implant site erosion (General disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram change (Investigations) | 0 (0) | 0 (0) | 1 (1)
Electroencephalogram abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Anastomotic stenosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Cardiac valve replacement complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Device malfunction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Extrusion of device (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Multiple drug overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Postoperative ileus (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Renal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Intestinal adhesion lysis (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized Cohort: InterStim Therapy Group (N=51) | Randomized Cohort: Standard Medical Therapy Group (N=75) | All Implanted Cohort (N=272)
Urinary tract infection (Infections and infestations) | 11 (14) | 3 (3) | 74 (123)
Undesirable change in stimulation (General disorders) | 6 (8) | 0 (0) | 60 (75)
Implant site pain (General disorders) | 3 (3) | 0 (0) | 40 (55)
Nasopharyngitis (Infections and infestations) | 4 (4) | 2 (2) | 15 (18)
Sinusitis (Infections and infestations) | 4 (4) | 2 (2) | 21 (28)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 33 (39)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 2 (2) | 26 (34)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 4 (4) | 5 (5)
Drug toxicity (Injury, poisoning and procedural complications) | 0 (0) | 7 (7) | 13 (18)
Constipation (Gastrointestinal disorders) | 1 (1) | 7 (7) | 19 (25)
Therapeutic product ineffective (General disorders) | 0 (0) | 0 (0) | 37 (42)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 27 (31)
Depression (Psychiatric disorders) | 2 (2) | 1 (1) | 27 (30)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 25 (27)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 22 (25)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 21 (28)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 19 (25)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 19 (22)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 19 (19)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 18 (19)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 17 (19)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 17 (17)
Cystitis interstitial (Renal and urinary disorders) | 0 (0) | 0 (0) | 16 (23)
Stress incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 16 (17)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 15 (15)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 15 (19)
Lead migration/dislodgment (General disorders) | 2 (2) | 0 (0) | 14 (17)

LIMITATIONS AND CAVEATS:
Predominantly female and Caucasian subjects could detract from generalizability. Centers followed individual protocols for peri-op antibiotics, lead choice, and procedure techniques. Lack of standardization may have impacted overall study results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No